CLINICAL TRIAL: NCT06939452
Title: A Single-arm, Multicenter Exploratory Clinical Trial of Anlotinib Combined With TQB2450 and the SOX Regimen as First-line Treatment for Advanced Gastric Cancer With Low PD-L1 Expression
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yongxu Jia (Other)
Responsible Party: Sponsor-Investigator, Yongxu Jia, Doctor, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMMUNOVA
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-03

CONDITIONS: Advanced Gastric or Gastroesophageal Junction (G/GEJ) Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- anlotinib +TQB2450 + Oxaliplatin+S-1 (Experimental)
  Interventions: Drug: anlotinib +TQB2450 + Oxaliplatin+S-1

INTERVENTIONS:
Drug: anlotinib +TQB2450 + Oxaliplatin+S-1 — Anlotinib: 10mg, po, d1-14,q3w,until disease progression or unacceptable toxicity.
  TQB2450: 1200mg, iv, d1, q3w,until disease progression or unacceptable toxicity. Oxaliplatin: 130mg/㎡, iv, d1,6 cycles.
  S-1:40mg, po, bid, d1~14,6 cycles.

SUMMARY:
To evaluate the efficacy and safety of anlotinib combined with TQB2450 and the SOX regimen as first-line treatment for advanced gastric cancer with low PD-L1 expression

DETAILED DESCRIPTION:
Evaluation of the efficacy and safety of anlotinib in combination with TQB2450 and the SOX regimen as first-line treatment for advanced gastric cancer with low PD-L1 expression. Additionally, real-world data were collected from hospital-based patients receiving immune checkpoint inhibitor (ICI)-combined chemotherapy as first-line therapy for PD-L1-low advanced gastric cancer to establish an external control cohort. The efficacy outcomes between the two treatment strategies were then compared.

ELIGIBILITY:
Inclusion Criteria:

* 1. Willing and able to provide written informed consent and comply with study procedures.
* 2. Histologically or cytologically confirmed HER2-negative (or HER2 status undetermined) unresectable locally advanced or metastatic gastric/gastroesophageal junction adenocarcinoma (including signet ring cell carcinoma, mucinous adenocarcinoma, and hepatoid adenocarcinoma variants).
* 3. Disease recurrence >6 months after completion of (neo)adjuvant chemotherapy or radiotherapy.
* 4. At least one measurable or evaluable lesion according to RECIST v1.1 criteria. Measurable lesions must not have received prior local therapy (e.g., radiotherapy); however, lesions within previously irradiated fields may be designated as target lesions if documented progression is demonstrated per RECIST v1.1.
* 5. Age 18-75 years.
* 6. ECOG performance status 0-1.
* 7. Life expectancy ≥3 months.
* 8. Organ Function Requirements and Laboratory Test Criteria During Screening (1) Complete Blood Count (CBC) Criteria： Hemoglobin (Hb): ≥ 90 g/L (no blood transfusion within 14 days) Absolute Neutrophil Count (ANC): ≥ 1.5 × 10⁹/L Platelet Count (PLT): ≥ 100 × 10⁹/L (no use of interleukin-11 [IL-11] or thrombopoietin [TPO] within 14 days) White Blood Cell Count (WBC): ≥ 4.0 × 10⁹/L (no granulocyte colony-stimulating factor [G-CSF] administration within 14 days) (2) Biochemical Panel Requirements: Total Bilirubin (TBIL): ≤ 1.5 × ULN (upper limit of normal),Alanine Aminotransferase (ALT) & Aspartate Aminotransferase (AST): ≤ 2.5 × ULN,Serum Creatinine (Cr): ≤ 1.5 × ULN or Creatinine Clearance (CrCl): ≥ 60 mL/min (calculated by Cockcroft-Gault formula),Serum Albumin: ≥ 25 g/L (2.5 g/dL) For Subjects with Hepatic Metastases:Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT): ≤ 5 × ULN，White Blood Cell Count (WBC): ≥ 4 × 10⁹/L，Platelet Count (PLT): ≥ 100 × 10⁹/L (without transfusion support)， Absolute Neutrophil Count (ANC): ≥ 1.5 × 10⁹/L (without granulocyte colony-stimulating factor [G-CSF] therapy) (3) Cardiac Function Assessment (Echocardiography)：Left Ventricular Ejection Fraction (LVEF): ≥ 50% (or above institutional lower limit of normal) (4) Coagulation Profile：International Normalized Ratio (INR) or Prothrombin Time (PT): ≤ 1.5 × ULN
* 9. Women of reproductive age must use effective contraception during the study period, after the last dose, and for at least 6 months following chemotherapy. It is recommended to start using contraception at least 3 months before the administration of the investigational drug; unsterilized males must also be required to use effective contraception for at least 6 months during the study period, after the last dose, and following chemotherapy. It is recommended to start using contraception at least 3 months before the administration of the investigational drug.
* 10. PD-L1 combined positive score ( CPS) <5

Exclusion Criteria:

* 1. Prior treatment with anlotinib hydrochloride or any immune checkpoint inhibitors (anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibodies);
* 2. History of immunodeficiency disorders, including HIV infection, other acquired or congenital immunodeficiency diseases, or prior organ transplantation;
* 3. Active hepatitis B or C infection, or active pulmonary tuberculosis;
* 4. CT-confirmed ulcerative lesions or fecal occult blood positivity;
* 5. History of clinically significant bleeding (excluding epistaxis) within 1 month prior to enrollment;
* 6. Previous allogeneic bone marrow or solid organ transplantation;
* 7. Interstitial lung disease including idiopathic pulmonary fibrosis, drug-induced pneumonitis, organizing pneumonia, or CT-confirmed active pneumonia;
* 8. Administration of live attenuated vaccines within 4 weeks before study initiation or anticipated during the study through 5 months post-treatment;
* 9. Systemic corticosteroids (>10 mg/day prednisone equivalent) or immunosuppressive therapy within 2 weeks prior to study initiation (inhaled or topical corticosteroids are permitted);
* 10. Known symptomatic CNS metastases or leptomeningeal carcinomatosis. Patients with previously treated CNS metastases may be eligible if neurologically stable for ≥4 weeks without steroids or anticonvulsants;
* 11. Conditions impairing oral drug absorption (e.g., dysphagia, chronic diarrhea, or intestinal obstruction);
* 12. Grade ≥2 peripheral neuropathy per NCI CTCAE v5.0;
* 13. Active infections requiring systemic antibiotics within 14 days prior to study entry;
* 14. Hepatic tumor burden exceeding 50% of total liver volume;
* 15. Bone metastases with impending spinal cord compression risk;
* 16. Uncontrolled comorbidities including:
* Poorly controlled hypertension (SBP ≥150 mmHg or DBP ≥100 mmHg despite antihypertensives)
* Grade ≥2 myocardial ischemia, myocardial infarction, or arrhythmias (QTc ≥480 ms)
* NYHA Class III-IV heart failure or LVEF <50% by echocardiography
* Uncontrolled active infections
* Decompensated liver cirrhosis or active hepatitis
* Uncontrolled diabetes (FBG >10 mmol/L)
* Proteinuria ≥++ on dipstick or confirmed 24-hour urinary protein >1.0 g
* 17. Non-healing wounds or fractures;
* 18. Coagulopathy (INR >1.5 or aPTT >1.5×ULN), bleeding diathesis, or requiring therapeutic anticoagulation:
* Known bleeding disorders (hemophilia, coagulopathies) or thrombocytopenia
* Hemoptysis (>2.5 mL/day) within 2 months
* Clinically significant bleeding within 3 months (GI bleeding, hemorrhagic ulcers, etc.)
* Chronic anticoagulation (warfarin/heparin) or antiplatelet therapy (aspirin ≥300 mg/day or clopidogrel ≥75 mg/day)
* 19. Major surgical procedures within 4 weeks prior to study or anticipated during treatment;
* 20. History within 6 months of:
* GI perforation/fistula
* Arterial/venous thromboembolism (excluding stable cerebral infarcts)
* 21. Clinically significant pleural/peritoneal effusions requiring intervention (asymptomatic minimal effusions not requiring treatment may be permitted);
* 22. Severe malnutrition;
* 23. Active substance abuse or psychiatric disorders impairing compliance;
* 24. Other active malignancies except:
* Curatively treated malignancies with >2 year disease-free interval
* Adequately treated non-melanoma skin cancer or lentigo maligna
* Carcinoma in situ with complete resection
* 25. Pregnancy or lactation;
* 26. Any condition deemed by investigators to compromise patient safety or study integrity;
* 27. Participation in other clinical trials within 30 days prior to enrollment or planned during study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2025-06-07 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | about 2 years
  The RECIST1.1 standards were used to evaluate the efficacy of drugs.

SECONDARY OUTCOMES:
Disease Control Rate(DCR) | about 2 years
Progression Free Survival(PFS) | about 2 years
Duration of Response(DOR) | about 2 years
1-year OS rate | about 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yongxu Jia, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided